CLINICAL TRIAL: NCT03153059
Title: The Association Between Gut Microbiota and Stool Frequency
Brief Title: Gut Microbiota and Stool Frequency
Status: Completed | Type: Observational
Sponsor: Kosin University Gospel Hospital (Other)
Responsible Party: Principal Investigator, Jae Hyun Kim, The association between gut microbiota and stool frequency, Kosin University Gospel Hospital
Other Study IDs: 2017-02-017-001
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Gut Microbiota
Keywords: gut microbiota; stool frequency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect the stool from participants, and extract DNA from stool sample. We plan to acquire the Human Derivative Research Description.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: a large number of defecation group (≥ 2-3 times/day) - 20 subjects
  Interventions: Other: Stool frequency
- group 2: normal defecation group (1 time/day or 1 time/2 days) - 20 subjects
  Interventions: Other: Stool frequency
- group 3: a small number of defecation group (≤ 2 times/week) - 20 subjects
  Interventions: Other: Stool frequency

INTERVENTIONS:
Other: Stool frequency — This study is just observational study.

SUMMARY:
We hypothesized that some difference in the composition and distribution of gut microbiota in people with a large number of defecation (two or three times a day or more), people with normal defecation (one time a day or two days), and people with a small number of defecation (two times a week or less).

And we investigate the association between gut microbiota and stool frequency.

DETAILED DESCRIPTION:
We divided three groups. (total number = 60 subjects)

1. a large number of defecation group (≥ 2-3 times/day) - 20 subjects
2. normal defecation group (1 time/day or 1 time/2 days) - 20 subjects
3. a small number of defecation group (≤ 2 times/week) - 20 subjects

After collection of stools, we will analyze the composition and distribution of gut microbiota, and compared the results of three groups.

ELIGIBILITY:
Inclusion Criteria:

* adults between the age of 20 and 50

Exclusion Criteria:

* subjects with cancer or IBD (inflammatory bowel disease)
* subjects with history of abdominal surgery
* subjects who take medication related to gastrointestinal motility within 3 months
* subjects who take antibiotics within 3 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
stool frequency and gut microbiota | six months
  Analysis of correlation between stool frequency and gut microbiota

SECONDARY OUTCOMES:
stool consistency and gut microbiota | six months
  Analysis of correlation between stool consistency and gut microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- Kosin University Gospel Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No
We have no plan to share IPD to other researchers.